CLINICAL TRIAL: NCT01224821
Title: Multicenter, Phase II Dosimetry/Validation Study of 131Iodine-Anti B1 (Murine) Radioimmunotherapy for Chemotherapy Refractory Low Grade B Cell Lymphomas and Low Grade Lymphomas That Have Transformed to Higher Grade Histologies
Brief Title: Dosimetry/Validation Study of 131Iodine-Anti B1 (Murine) Radioimmunotherapy for Chemotherapy Refractory Low Grade B Cell Lymphomas and Low Grade Lymphomas That Have Transformed to Higher Grade Histologies
Acronym: RIT-II-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104731
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: iodine I 131 tositumomab; anti-B1 Antibody; Bexxar; radioimmunotherapy; tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- Tositumomab and Iodine I-131 Tositumomab (Experimental): Patients receive a dosimetric dose consisting of 450 milligrams (mg) of unlabeled tositumomab (TST, Anti-B1 Antibody) intravenously (IV) followed by 5 milliCurie (mCi) of Iodine I 131 TST IV. Serial whole body sodium iodide probe scintillation counts and whole body conjugate view gamma camera scans obtained approximately 1 hour after administration and then daily for the next 7 days were used to determine the radioactive clearance and the dose of iodine I 131 TST required to deliver a 75 centigray (cGy) therapeutic dose. The therapeutic dose was administered 7-14 days after the dosimetric dose and consisted of TST 450 mg and an activity of Iodine 131 calculated to deliver 75 cGy or 65 cGy of total body irradiation, depending on platelet count, and 35 mg TST.
  Interventions: Biological: Tositumomab (Anti-B1 Antibody) and Iodine-131 Tositumomab

INTERVENTIONS:
Biological: Tositumomab (Anti-B1 Antibody) and Iodine-131 Tositumomab — Patients receive a dosimetric dose consisting of 450 milligrams (mg) of unlabeled tositumomab (TST, Anti-B1 Antibody) intravenously (IV) followed by 5 milliCurie (mCi) of Iodine I 131 TST IV. Serial whole body sodium iodide probe scintillation counts and whole body conjugate view gamma camera scans obtained approximately 1 hour after administration and then daily for the next 7 days were used to determine the radioactive clearance and the dose of iodine I 131 TST required to deliver a 75 centigray (cGy) therapeutic dose. The therapeutic dose was administered 7-14 days after the dosimetric dose and consisted of TST 450 mg and an activity of Iodine 131 calculated to deliver 75 cGy or 65 cGy of total body irradiation, depending on platelet count, and 35 mg TST.

SUMMARY:
Study RIT-II-001 is a phase II, multicenter study of the safety, tumor and organ dosimetry, dosimetry methods, and efficacy of Iodine-131 Anti-B1 Antibody for the treatment of patients with low-grade or transformed low-grade non-Hodgkin's lymphoma (NHL). The primary objective of this study is to demonstrate that each site could accurately conduct the whole body dosimetry required for the safe and effective dosing of Iodine-131 Anti-B1 Antibody. Additional objectives of this study are to evaluate the efficacy, dosimetry, and safety of Iodine-131 Anti-B1 Antibody.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a histologically confirmed diagnosis of low-grade non-Hodgkin's B-cell lymphoma or low-grade lymphoma that has transformed to intermediate-, or high-grade lymphoma (transformed lymphoma) according to the Working Formulation for Clinical Usage (IWF A, B, and C).
* Patients must have evidence that their tumor tissue expresses the CD20 antigen.
* Patients must have progressive disease of either low-grade or transformed lymphoma within one year of completion of the last chemotherapy regimen administered.
* Patients must have been previously treated with at least one chemotherapy regimen that included an anthracycline or anthracenedione.
* Patients must have a performance status of at least 60% on the Karnofsky Scale and anticipated survival of at least three months.
* Patients must have an absolute granulocyte count of over 1,500 /mm3 and a platelet count above 100,000 /mm3 within seven days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have normal renal function (creatinine less than 2.0 mg/dL) and hepatic function (bilirubin less than 2.0 mg/dL) within seven days of study entry.
* Patients must have bi-dimensionally measurable or evaluable progressive lymphoma disease (at least a 25% increase in tumor size or new sites of disease when compared to the last best disease response). Progression must have occurred within 12 months of the preceding response.
* Patients must be at least 18 years of age.
* Patients must give written informed consent and sign an approved informed consent form prior to study entry.

Exclusion Criteria

* Patients with more than an average of 25% of the intertrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically at study entry.
* Patients who have received cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within FOUR weeks prior to study entry (six weeks for nitrosourea compounds) or who exhibit persistent clinical evidence of toxicity. The use of steroids must have been discontinued (except maintenance-dose steroids) at least one week prior to study entry and patients must then show evidence of stable or progressive disease.
* Patients with prior hematologic stem cell transplant following high-dose chemotherapy or chemo/radiotherapy .
* Patients with obstructive hydronephrosis.
* Patients with evidence of active infection requiring intravenous antibiotics at the time of study entry.
* Patients with New York Heart Association class 3 or 4 heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which patient has been disease-free for five years.
* Patients with known HIV infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant. Patients of child-bearing potential must undergo a pregnancy test within seven days of study entry. Males and females must agree to use effective contraception during the study.
* Patients with previous allergic reactions to iodine. This does not include IV contrast materials.
* Patients who were previously given any monoclonal or polyclonal antibodies of any foreign species for either diagnostic or therapeutic purposes. This includes engineered chimeric and humanized antibodies.
* Patients who previously received radioimmunotherapy.
* Patients with progressive disease in a field that has been previously irradiated with more than 3500 cGy.
* Patients who are on another protocol involving non-approved drugs or biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 1995-12; Primary Completion 1997-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) received radioimmunotherapy of tositumomab (TST) and Iodine I 131 TST in 2 phases (Ph.): Ph. 1, dosimetric dose; Ph. 2, therapeutic dose. Par. were evaluated until disease progression, they died, or they were on study for 2 years. Par. completing 2 years of study could enter a long-term follow-up study (BEX104526; NCT00240591).
Groups:
- TST and Iodine I 131 TST: Participants received a dosimetric dose (DD) consisting of 450 milligrams (mg) of unlabeled tositumomab (TST) intravenously (IV) followed by 5 milliCurie (mCi) of Iodine I 131 TST IV. Serial whole body sodium iodide probe scintillation counts and whole body conjugate view gamma camera scans obtained approximately 1 hour after DD administration and then daily for the next 7 days were used to determine the radioactive clearance (RC) and the dose of iodine I 131 TST required to deliver a 75 centigray (cGy) therapeutic dose (TD). The TD was administered 7-14 days after the DD and consisted of TST 450 mg and an activity of Iodine 131 calculated to deliver 75 cGy or 65 cGy of total body irradiation, depending on platelet count, and 35 mg TST. Participants who had completed at least 6 months of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in Study BEX104526 were followed for up to 10 years.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and Iodine I 131 TST
Started | 47
Completed | 1 (This participant completed the study per Protocol Amendment 2.)
Not Completed | 46
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 38
Not completed — Continued Follow-up in Study BEX104526 | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Started Other Treatment | 1
Period: Long-Term Follow-Up
Arm/Group | TST and Iodine I 131 TST
Started | 11 (11/47 participants withdrawing from this study enrolled in the LTFU study for continued evaluation.)
Completed | 0
Not Completed | 11
Not completed — Death | 2
Not completed — Completion of 10 Year Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (12)
Gender [Count of Participants; unit: Participants]
  Female | 22
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45
  Asian | 1
  Black | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received the Therapeutic Dose at the Seven Clinical Research Sites
Description: The dosimetry methods were validated for seven different clinical research sites.
Time Frame: Day 1 within one hour of infusion (I) and prior to urination (U); Days 2, 3, and 4 after dosimetric dose (DD) I, following U; Days 6 and 7 after DD I, following U
Population: Intent-to-Treat (ITT) Exposed Population: all participants who enrolled in the study and received at least one dose of study drug. One participant did not receive the therapeutic dose.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 46
participants
  Clinical site 003 | 7
  Clinical site 004 | 8
  Clinical site 005 | 8
  Clinical site 006 | 5
  Clinical site 007 | 6
  Clinical site 008 | 6
  Clinical site 009 | 6

2. Secondary Outcome: Number of Participants With the Indicated Therapeutic Doses (TD) (Total Body Dose)
Description: Based on their platelet count and body weight. Participants received different TDs of TST. For obese participants (weighing more than 137% of their calculated lean body weight), the calculation to determine the administered activity (mCi) was performed using the maximum effective mass (i.e., the minimum of the participant's mass and 137% of their calculated lean body weight). The administered activity (mCi) for participants with a Baseline platelet count of 100001-149999 cells/millimeter cubed (mm^3) was reduced to a 65 cGy total body dose, after any adjustment for obesity.
Time Frame: Participants were evaluated for up to 142 months in Study 104731 or were followed in the long-term follow-up study (Study 104526) for up to 136.3 months
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 47
participants
  0 cGy | 1
  53 cGy | 1
  65 cGy | 9
  75 cGy | 36

3. Secondary Outcome: Number of Participants (Par.) With Response (CR, CCR, or PR), as Assessed by the Investigator
Description: Par. with response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 46
participants | 27

4. Secondary Outcome: Number of Participants With Confirmed Response (CR, CCR, or PR), as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 39
participants | 23

5. Secondary Outcome: Number of Participants With CR and CCR, as Assessed by the Investigator
Description: The total number of participants with CR and CCR was reported. CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. Clinical Complete Response: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 46
participants | 15

6. Secondary Outcome: Number of Participants With Confirmed CR and CCR, as Assessed by the Investigator
Description: The total number of participants with CR and CCR was reported. Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. Clinical Complete Response: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants evaluable for confirmed CR and CCR were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 39
participants | 14

7. Secondary Outcome: Duration of Response for All Confirmed Responders (CR, CCR, or PR), as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Duration of response is defined as the time from the first documented response until disease progression. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 23
months | 14.3 [7.4 to 31.2]

8. Secondary Outcome: Duration of Response for All Unconfirmed Responders (CR, CCR, or PR), as Assessed by the Investigator
Description: Duration of response is defined as the time from the first documented response until disease progression. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 27
months | 9.9 [4.2 to 31.2]

9. Secondary Outcome: Duration of Response for All Confirmed Complete Responders, as Assessed by the Investigator
Description: as for outcome 7
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed CR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 11
months | 31.2 [13.6 to 95.9]

10. Secondary Outcome: Duration of Response for All Unconfirmed Complete Responders, as Assessed by the Investigator
Description: as for outcome 8
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed CR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 13
months | 31.2 [13.6 to 95.7]

11. Secondary Outcome: Duration of Response for All Confirmed Clinical Complete Responders, as Assessed by the Investigator
Description: as for outcome 7
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed CCR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 2
months | 17.2 [14.6 to 19.9]

12. Secondary Outcome: Duration of Response for All Unconfirmed Clinical Complete Responders, as Assessed by the Investigator
Description: as for outcome 8
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants with a confirmed CCR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 2
months | 17.2 [14.6 to 19.9]

13. Secondary Outcome: Median Time to Treatment Failure for All Participants
Description: Time to treatment failure is defined as the length of time from the date of enrollment to the first incidence of treatment withdrawal, study removal, progression, and/or alternative therapy for the participant's lymphoma, or death.
Time Frame: as for outcome 2
Population: ITT Exposed Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 47
months | 5 [3 to 7]

14. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause. Time to death is the time from the dosimetric dose to the date of death.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only those participants who died during the study were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 34
months | 35.3 [24.7 to 83.4]

15. Secondary Outcome: Time to Disease Progression or Death for Responders, as Assessed by the Investigator
Description: Progression-free survival or time to progression is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death.
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only participants classified as responders with disease progression or those who died were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 45
months | 5.3 [3.2 to 6.6]

16. Secondary Outcome: Time to Disease Progression or Death for All Participants, as Assessed by the Investigator
Description: as for outcome 15
Time Frame: as for outcome 2
Population: ITT Exposed Population. Only participants with disease progression or those who died were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 47
months | 5 [3 to 7]

ADVERSE EVENTS:
Arm/Group | TST and Iodine I 131 TST
Serious Adverse Events (participants affected / at risk) | 23/47
Other Adverse Events (participants affected / at risk) | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=47)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or Oral Cavity Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bacteremia (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Device Related Sepsis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Pneumococcal Sepsis (Infections and infestations) | 1
Staphylococcal Sepsis (Infections and infestations) | 1
Urinary Tract Infection Enterococcal (Infections and infestations) | 1
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Multi-Organ Failure (General disorders) | 1
Hypotension (Vascular disorders) | 3
Orthostatic Hypotension (Vascular disorders) | 1
Serum Sickness (Immune system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=47)
Fatigue (General disorders) | 19
Pyrexia (General disorders) | 16
Edema Peripheral (General disorders) | 6
Chills (General disorders) | 5
Local Swelling (General disorders) | 2
Mucous Membrane Disorder (General disorders) | 2
Asthenia (General disorders) | 1
Catheter Site Erythema (General disorders) | 1
Catheter Site Pain (General disorders) | 1
Chest Discomfort (General disorders) | 1
Extravasation (General disorders) | 1
Feeling Abnormal (General disorders) | 1
Gait Disturbance (General disorders) | 1
Hunger (General disorders) | 1
Infusion Site Extravasation (General disorders) | 1
Localized Edema (General disorders) | 1
Malaise (General disorders) | 1
Multi-Organ Failure (General disorders) | 1
Absolute Neutrophill Count (ANC) <1000 cells/cubic millim(cm (Investigations) | 29
Platelets < 50,000 cells/cmm (Investigations) | 27
WBC (White Blood Cells) < 2,000 cells/cmm (Investigations) | 27
Hemoglobin < 8.0 grams/deciliter (g/dL) (Investigations) | 11
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 12
Abdominal Pain (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1
Abdominal Tenderness (Gastrointestinal disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal Reflux disease (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal Fissure (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5
Herpes Zoster (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Viral Infection (Infections and infestations) | 2
Bacteremia (Infections and infestations) | 1
Bacterial Infection (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Device Related Sepsis (Infections and infestations) | 1
Herpes Virus Infection (Infections and infestations) | 1
Infusion Site Cellulitis (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pneumococcal Sepsis (Infections and infestations) | 1
Pseudomonas Infection (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Staphylococcal Sepsis (Infections and infestations) | 1
Urinary Tract Infection Enterococcal (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Ageusia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Post Herpetic Neuralgia (Nervous system disorders) | 1
Sensory Disturbance (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Choking Sensation (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Blistering (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2
Blood Blister (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Anemia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypothyroidism (Endocrine disorders) | 9
Hypotension (Vascular disorders) | 4
Flushing (Vascular disorders) | 2
Orthostatic Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Ear Discomfort (Ear and labyrinth disorders) | 1
Serum Sickness (Immune system disorders) | 2
Anaphylactic Reaction (Immune system disorders) | 1
Weight Decreased (Investigations) | 2
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1
Oliguria (Renal and urinary disorders) | 1
Ureteric Obstruction (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Conjunctivitis (Eye disorders) | 1
Periorbital Edema (Eye disorders) | 1
Confusional State (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Vaginal Lesion (Reproductive system and breast disorders) | 1
Tachycardia (Cardiac disorders) | 1
Spinocerebellar Ataxia (Congenital, familial and genetic disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.